CLINICAL TRIAL: NCT04586881
Title: Catch me if You Can - the Individual Relationship Between Potential Ablation Targets From CARTOFINDER and Myocardial Fibrosis
Status: Completed | Type: Observational
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HDZ_ER001_CS
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Single center observational study to compare the relationship between atrial fibrosis and potential ablation targets from CARTOFINDER.

DETAILED DESCRIPTION:
A total number of 30 patients will undergo catheter Ablation for persistent AF. Pre-procedural cardiac MRI will be performed with late-gadolinium enhancement to visualize the individual amount and distribution of fibrosis in the right and left atrium. CARTOFINDER-guided mapping will be performed during the ablation procedure followed by AF ablation. The individual relationship between atrial fibrosis and potential ablation targets will be accessed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing their 1st AF ablation procedure for persistent atrial fibrillation (AF) as per recent Heart Rhythm Society (HRS) consensus document
2. Able to understand and willing to sign the Informed Consent Form.
3. Age ≥18 years.

Exclusion Criteria:

1. Contraindication for DE-MRI with a full dose of Gadolinium-based contrast agent.
2. Previous left atrial ablation or surgical procedure
3. Renal failure with CrCl <60 ml/min
4. Women currently pregnant, breastfeeding, or of childbearing age not currently taking or not willing to use a reliable form of contraception
5. Mental or physical inability to take part in the study
6. Uncontrolled hypertension
7. Morbid obesity (BMI > 35), or inability to be placed in MRI due to body mass.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 20 consecutive patients with drug-refractory persistent AF will be included in this prospective observational analysis. AF will be defined as persistent if episodes lasted > 7 days or required electrical or pharmacological cardioversion after ≥ 48 h from onset. All patients will be treated for AF at the Heart and Diabetes Center NRW, Bad Oeynhausen, Germany. Written informed will be obtained from each patient, the study concept complies with the Declaration of Helsinki and the institutional review board already approved the study design. Catheter ablation will be performed under deep sedation. In all patients preprocedural Magnetic Resonance Imaging (MRI) will be performed to guide the intervention, visualize the individual amount and distribution of fibrosis and to visualize the anatomical location and course of the esophagus.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
AF recurrence | 12 months
  recurrence of atrial fibrillation after catheter ablation

CONTACTS AND LOCATIONS:
Locations (1):
- Herz- und Diabeteszentrum NRW, Ruhr-Universität Bochum, Bad Oeynhausen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guckel D, Piran M, Bergau L, Hamriti ME, Fink T, Sciacca V, Reil JC, Braun M, Khalaph M, Imnadze G, Kramer K, Friedrich S, Ruhl J, Korperich H, Sommer P, Sohns C. The individual relationship between atrial fibrillation sources from CARTOFINDER mapping and atrial cardiomyopathy: The catch me if you can trial. Pacing Clin Electrophysiol. 2023 Dec;46(12):1553-1564. doi: 10.1111/pace.14847. Epub 2023 Oct 27. PMID 37885302